CLINICAL TRIAL: NCT06158698
Title: Single-blinded Randomized Investigator-initiated Controlled Trial to Assess the Efficacy of Colchicine to Treat Patients With Cardiomyopathy With Myocarditis (Chronic Inflammatory Cardiomyopathy)
Brief Title: CMP-MYTHiC Trial and Registry - CardioMyoPathy With MYocarditis THerapy With Colchicine
Acronym: CMP-MYTHiC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Niguarda Hospital (Other)
Collaborators: European Union (Other); Ministry of Health, Italy (Other Government); Mario Negri Institute for Pharmacological Research (Other); University of Milano Bicocca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMP-MYTHiC; PNRR-MAD-2022-12376225 (Other Grant/Funding Number: European Union- NextGenerationEU)
Record Dates: First submitted 2023-11-15; First posted 2023-12-06 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Cardiomyopathies; Myocarditis; Inflammatory Cardiomyopathy; Heart Failure; Ventricular Arrythmia
Keywords: treatment; trial; colchicine; registry; inflammation; outcome; genetic testing
MeSH Terms: conditions — Cardiomyopathies; Myocarditis; Heart Failure; Inflammation | interventions — Colchicine; Therapeutics

STUDY DESIGN:
Intervention Model Description: Two-parallel groups randomized, single-blinded, multi-center phase III-controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colchicine (Experimental): Patients treated with colchicine 0.5-1 mg (1 mg if tolerated) for 6 months.
  Interventions: Drug: Colchicine
- Placebo (Placebo Comparator): Patients treated with placebo tablets.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Colchicine — Colchicine 1 mg daily (or 0.5 mg daily il weight <70 kg) from randomization for 180 days (6 months)
  Other Names: Treatment
  Arms: Colchicine
Other: Placebo — Placebo 1 mg daily (or 0.5 mg daily il weight <70 kg) from randomization for 180 days (6 months)
  Arms: Placebo

SUMMARY:
Two-parallel groups randomized, single-blinded, multi-center phase III controlled trial in patients with chronic inflammatory cardiomyopathy to assess the efficacy of colchicine and associated prospective registry to assess the prognostic value of positive genetic testing in this population.

DETAILED DESCRIPTION:
In a proportion of patients, myocarditis, an inflammatory injury of cardiomyocytes (CMs), can lead to chronic inflammatory cardiomyopathy (Infl-CMP) characterized by an increased risk of life-threatening ventricular arrhythmias (VA) or ventricular dysfunction and heart failure (HF). Most cases of myocarditis have a viral trigger or an autoimmune etiology, while genetic predisposition has been sporadically reported. Recent data point to a relevant role of genetics, with pathogenic genetic variants associated with dilated or arrhythmic cardiomyopathies found in 8-31% of patients with Infl-CMP and left ventricular (LV) systolic dysfunction. Occasionally, patients with myocarditis may have a positive family history of cardiomyopathy, or sudden cardiac death (SCD), which can lead to genetic testing for myopathic cardiac gene variants (MCGV). Small series showed the co-existence of myocarditis and MCGV in patients with dilated cardiomyopathy. In this complex background, it is still unclear whether targeting myocardial inflammation with immunomodulating drugs can ameliorate the outcome of these patients.

TRIAL - The Investigators will conduct a Trial to assess whether in patients with Infl-CMP with VA or HF phenotype, colchicine compared with placebo can reduce myocardial inflammation improving the clinical condition of patients. In the trial both patients with positive MCGV and negative MCGV will be randomized, and the investigators check if the genetic background can affect the response to colchicine. The target of this pilot trial is to randomize 40 patients in each arm and have ideally 15 patients with MCGV(+) in each arm. The use of colchicine in our proposal of trial relies on the safety of colchicine, and the relatively low rate of side effects at low dosages. It has shown that colchicine performs its functions by inhibiting the activation of pore formation carried out by P2X2 and P2X7 receptors, that concur to the activation of the inflammasome, thus potentially targeting a specific cause observed in Infl-CMP.

In a pilot, randomized, and single-blinded trial the investigators look at the immunomodulating effect of colchicine 0.5-1 mg vs. placebo in patients with Infl-CMP based on cardiac magnetic resonance imaging (CMRI) or fluorodeoxyglucose (FGD)-positron emission tomography (PET) scan with VA (including high premature ventricular complexes [PVC] burden), reduced LV ejection fraction (EF), or significantly increased levels of natriuretic peptides but without indication to immunosuppression (i.e., associated systemic autoimmune disorders) to assess whether colchicine can improve myocardial inflammation or decrease troponin release or the burden of PVCs or improve the clinical outcome (major VA, HF hospitalizations). The duration of the trial will be 6 months. The rationale of the pilot (CMP-MYTHiC CardioMyoPathy with MYocarditis THerapy with Colchicine) trial is based on a recent registry of 55 symptomatic patients with >5000 premature ventricular complexes (PVCs)/24 hours with FDG-PET imaging consistent with Infl-CMP, where a signal of benefit was observed in patients who received prednisone 40 mg for 3 months. The benefit was defined as a reduction in the PVC burden >80% and negative FDG-PET scan at follow-up. It must be noted that up to 24% of these cases had a diagnosis of sarcoidosis, where there is already an indication to therapy with steroids. In this study (MAVERIC registry) the improvement of patients treated with prednisone alone was 84% vs. 33% in patients not taking prednisone. As the investigators expect a lower effect of colchicine compared with prednisone but with a safer drug profile than prednisone, the investigators considered a theoretical optimal response in patients taking colchicine of 66%, while the investigators expected a similar optimal response in patients taking placebo as in the MAVERIC registry in patients not taking prednisone. Thus, considering an increase in the probability to reach the primary endpoint, defined as proportion of patients that are alive and free of any worsening (clinical, arrhythmic burden and imaging outcome) and that shows at least one of the signs of improvements (IMAGING or ARRHYTMIC improvements) at 6 months from 33% in the placebo arm to 66% in the colchicine therapy arm, the planned sample size of 80 patients (40 per group) will allow achieving a power of 0.80 with an overall type I error of 0.025 using one-sided Fisher's Exact test.

Endpoints will be analyzed according to the following principles:

1. Intention-to-treat (ITT) population: patients according to assigned randomized treatment arm.
2. Per Protocol (PP) population: only patients allocated to the colchicine therapy arm who took the drug for at least 4 months will be considered in the experimental group. Patients assigned to the colchicine therapy arm that will receive less than 4-month colchicine therapy will be excluded from this population. Likely, patients allocated to the optimal medical therapy with placebo will be included if they have taken the placebo therapy for at least 4 months. Patients allocated to the treatment or placebo that will receive any immunosuppressive agents (e.g. corticosteroids) for at least 1 month during the trial will be excluded from this population.
3. A sensitivity analysis will also be performed on the previously defined populations after excluding patients (1) with an implantable cardioverter defibrillator (ICD) before randomization (2) who underwent a ventricular ablation before randomization (3) who were diagnosed with a systemic autoimmune disorder or a histological diagnosis of eosinophilic myocarditis, cardiac sarcoidosis or giant cell myocarditis after the randomization.

REGISTRY - The main aim is to determine if patients with positive MCGV (+) Infl-CMP have a worse outcome compared with patients with negative MCGV (-) Infl-CMP in terms of recurrence of VA, including a high burden of PVCs or HF episodes or reduced improvement of ventricular function or persistence of myocardial inflammation on follow-up CMRI or FDG-PET. Furthermore, the investigators investigated characteristics that can help to identify patients with likely positive genetic tests among patients presenting with Infl-CMP, and variables that are independently associated with prognosis in patients with Infl-CMP. If patients have criteria to enter the registry, but not the trial, or (2) if do not consent to be randomized while they are willing to be followed in the registry, or (3) if the number of 80 patients is reached in the trial, even if the patients have the criteria to be included in the trial, these patients will enter the prospective registry. The foreseen number of the patients in the registry is 50-70 during the study period. To reach the objectives of the registry, deep phenotypical characterization of patients presenting with chronic Infl-CMP with VA and HF phenotypes will be performed in association with genetic testing.

TRANSLATIONAL STUDY - the investigators will perform translational experiments from the blood sample and endomyocardial biopsy (EMB) from patients recruited in the trial and the registry, if they consent. In particular, 50 patients (the first 25 with positive genetics and 25 with negative genetics) who agree to donate 18 mL of their blood will enter the translational study. From the blood, the investigators will get human-induced pluripotent stem cells (iPSC-CM) to unveil the molecular mechanisms that are responsible for the inflammatory response in the myocardium. As a control group, the investigators will involve the first 25 family members of the probands with the negative cardiac phenotype (FMPNCP) test that agree to be sampled for the same amount of blood. The hypothesis of these experiments is that a specific genetic background identified in patients with Inf-CMP is sufficient to induce an inflammatory myocardial response. Briefly, the investigators will generate tridimensional cardiac tissues (EHTs) using CMs derived from human-iPSC-CM from patients with MCGV(+) Infl-CMP versus MCGV(-) Infl- CMP and FMPNCP. EHTs and CMs will be subjected to specific mechanical, cellular, and pharmacological stimuli to unveil the molecular mechanisms that are responsible for the inflammatory response. The results of these experiments, together with the molecular analysis of EMBs could reveal novel molecular pathways that will be relevant to specific personalized therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria Trial and Registry:

* Males and females with Infl-CMP associated with VA (including high PVC burden), reduced LVEF, or significantly increased levels of natriuretic peptides.
* Patients of 18 years or older
* Evidence of myocardial inflammation on CMRI (using 2018 Lake Louis criteria) or FDG-PET performed in the 3 months before randomization to be included in the trial OR in the last 12 months before for the registry.
* Presence of any of the following characteristics and if symptoms have been present for more than 1 month:
* Mono-morphic or polymorphic PVC burden of ≥3000 in 24 hours, or NSVTs (defined as >3 more consecutive beat lasting <30 seconds) or evidence of sustained ventricular tachycardias (SVT).
* Reduced LVEF on echocardiogram (<50%) or on CMRI (<60%)-. Increased N-terminal pro-B-type natriuretic peptide (NT- proBNP) concentration of 1000 pg/mL or more, or a B-type natriuretic peptide (BNP) concentration of 200 pg/mL or more
* Persistence of increased high-sensitivity troponin levels above the upper reference limit (URL) after at least 2 months from the first assessment and at least a mono-morphic or polymorphic PVC burden of ≥1000 in 24 hours.

Exclusion Criteria Registry:

* Proven history of myocardial infarction with evidence of ischemic scar on echocardiogram or CMRI,
* Significant flow-limiting coronary artery disease (stenosis above 50%) on invasive coronary angiography or computed tomography (CT) coronary angiography,
* Cardiomyopathy attributed to toxins such as alcohol and illicit drugs, or to specific causes (i.e. amyloidosis or hypertrophic cardiomyopathy)
* Known systemic autoimmune disorder (the exception will be for patients with systemic autoimmune disease or isolated cardiac sarcoidosis with a family history of cardiomyopathy, myocarditis, or arrhythmias, where overlap between an autoimmune event and a genetic background can occur). These patients will undergo genetic tests. Patients with autoimmune systemic disorders and isolated cardiac sarcoidosis with positive genetic tests for MCVG will be included in the registry.
* Previous history of cardiac surgery for instance correction of congenital heart disease or a valve repair/replacement
* Known chronic infective disease, such as HIV infection or tuberculosis
* Participants involved in another clinical trial, defined by the participation in a clinical trial in which an investigational drug was administered in the 30 days prior to screening, or 5 half-lives of the study drug, whichever is longer;
* Any other significant disease or disorder which (expected life expectancy <12 months), in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial or the participant's ability to participate in the trial.

Exclusion Criteria Trial :

* Proven history of myocardial infarction with evidence of ischemic scar on echocardiogram or CMRI,
* Significant flow-limiting coronary artery disease (stenosis above 50%) on invasive coronary angiography or computed tomography (CT) coronary angiography,
* Cardiomyopathy attributed to toxins such as alcohol and illicit drugs, or to specific causes (i.e. amyloidosis or hypertrophic cardiomyopathy)
* Known systemic autoimmune disorder (the exception will be for patients with systemic autoimmune disease or isolated cardiac sarcoidosis with a family history of cardiomyopathy, myocarditis, or arrhythmias, where overlap between an autoimmune event and a genetic background can occur). These patients will undergo genetic tests. Patients with autoimmune systemic disorders and isolated cardiac sarcoidosis with positive genetic tests for MCVG will be included in the registry.
* Previous history of cardiac surgery for instance correction of congenital heart disease or a valve repair/replacement
* Known chronic infective disease, such as HIV infection or tuberculosis
* Participants involved in another clinical trial, defined by the participation in a clinical trial in which an investigational drug was administered in the 30 days prior to screening, or 5 half-lives of the study drug, whichever is longer;
* Any other significant disease or disorder which (expected life expectancy <12 months), in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial or the participant's ability to participate in the trial.
* Women with childbearing potential (this exclusion criterion is due to insufficient human information regarding the embryofoetal risk with colchicine)
* Current symptomatic atrial arrhythmias (including persistent atrial fibrillation) associated with LV dysfunction,
* Advance heart failure (NYHA III or need for inotropes including levosimendan), or recurrent VA despite previous catheter ablation,
* Known systemic autoimmune disorder or other conditions at the time of randomization where immunosuppression is assumed useful (i.e. cardiac sarcoidosis),
* Patients already on chronic immunosuppressive therapies (including colchicine) or in whom immunosuppressive therapy is deemed necessary
* Contraindication to colchicine, including allergies to this medication and its excipients (i.e., lactose and sucrose),
* Impaired renal function (eGFR<30 ml/min/1.73m2),
* Known history of hepatic cirrhosis or transaminase levels at baseline > x3-fold the URL
* Patients with peripheral eosinophilia (eosinophil count >10% of the leukocytes) or known hypereosinophilic syndrome at the time of randomization.
* Severe gastrointestinal insufficiency (for instance, malabsorption syndrome, severe chronic diarrhea)
* Women during breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2026-05-02 (Estimated); Study Completion 2028-05-02 (Estimated)

PRIMARY OUTCOMES:
Patients alive and free of any worsening features (clinical, arrhythmic burden and imaging outcome) AND that show at least one of the signs of improvements (IMAGING or ARRHYTMIC improvements). | 6 months from randomization
  Clinical worsening (at least one of the following):
  1. cardiac death
  2. hospitalization for worsening HF or arrhythmic events,
  3. Sustained ventricular tachycardia (SVT).
  Worsening arrhythmic burden:
  1. PVC burden increase of 50% on ECG ambulatory monitoring
  2. Increase in NSVT of 30% compared with baseline
  3. Any SVT.
Worsening imaging outcomes | 6 months from randomization
  1. Proportion of patients with LVEF reduction >10%on echo/CMRI,
  2. Proportion of patients with new areas of edema on CMRI or FDG-PET associated with an increase in the edema in the inflammatory lesion identified on baseline CMRI or FDG-PET.
  Improvement of imaging outcome:
  1. Proportion of patients with a reduction in edema on CMRI or FDG without new areas of edema AND normal high sensitivity troponin.
  2. Proportion of patients with disappearance of edema on CMRI OR NO FDG uptake on PET Improvement of arrhythmic outcome:
  1. Improvement of ARRHYTHMIC burden. Proportion of patients with a PVC burden reduction of 70% on the ECG ambulatory monitoring and no NSVT/SVT.

SECONDARY OUTCOMES:
LVEF change on echocardiogram. | 6 months from randomization
  Absolute change at 6 months from randomization of the LVEF on echocardiogram. Patients not performing echocardiography due to death, heart transplantation (HTx) will be counted as -10 point in the LVEF.
LVEF change on CMRI | 6 months from randomization
  Absolute change at 6 months from randomization of the LVEF on CMRI when available. Patients not performing the CMRI due to death, HTx, LVAD implantation or device implantation after randomization will be counted as -10 point in the LVEF.
Evidence of dysfunction and/or dilation on CMRI | 6 months from randomization
  Proportion of patients with LVEF<55% AND/OR LV dilation on 6-month CMRI (CMRI clips will be centrally reviewed) or not performing the CMRI due to death, HTx, LVAD implantation or device implantation after randomization (i.e. ICD).
Clinical secondary endpoints | 6 months from randomization
  Composite endpoint: (1) all-cause death or (2) HTx or (3) LVAD implantation, or (5) first rehospitalization due to HF or VA, or advanced atrioventricular (AV) block.
Mortality | 6 months from randomization
  All-cause deaths
Time to HF or arrhythmic events | 6 months from randomization
  Time to hospitalization for HF/VA or advanced AV block
Changes on ambulatory ECG monitoring | 6 months from randomization
  Composite endpoint of NSVT OR increased burden of PVCs (>5%) on 24-hour ECG ambulatory monitoring, performed at 6- months
Changes in Quality of life | 6 months from randomization
  Changes in quality of life at 6 months follow up compared with baseline using 2 different questionnaires: the EoQ-5D-5L and KCCQ (CSS and OSS)
Need for immunosuppression | 6 months from randomization
  Need to initiate an immunosuppressive drug

OTHER OUTCOMES:
The primary aim of the REGISTRY is the proportion of patients with MCGV(+) Infl-CMP versus MCGV(-) Infl-CMP with more primary endpoints | Minimum follow up at 6 months
  We will measure the outcome of the patients in the registry as described in the TRIAL at the end of a minimum follow-up of 6 months.
  The co-primary aim of the registry will be to the identify baseline variables that are independently associated with the above-mentioned 6-month endpoints.
  The patients who enter the registry are expected to follow an even longer follow-up of 2
  The Registry endpoints pooling together patients included in the trial and registry.
Differences in the results of in-vitro experiments between MCGV(+) vs. MCGV(-) Infl-CMP patients and between MCGV(+) Infl-CMP patients and family members of the probands with the negative cardiac phenotype (FMPNCP) | Minimum follow up at 6 months
  We will compare in-vitro experiments between MCGV(+) vs. Infl-CMP versus MCGV(-) Infl-CMP patients and between MCGV(+) Infl-CMP patients and family members of the probands with the negative cardiac phenotype (FMPNCP). Samples for the experiments will be from patients included in the trial and registry.

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Ammirati, MD, PhD, Principal Investigator — ASST Grande Ospedale Metropolitano Niguarda
Locations (10):
- Italy (10):
  - Università degli studi della Campania L.Vanvitelli e Azienda Ospedaliera Specialistica dei Colli - Ospedale Monaldi, Napoli, Campania
  - Policlinico S.Orsola-Malpighi, Bologna, Emilia-Romagna
  - Azienda Sanitaria Universitaria Integrata Giuliano Isontina, Trieste, Trieste, Friuli Venezia Giulia
  - Presidio Ospedaliero Universitario "Santa Maria della Misericordia", Udine, Friuli Venezia Giulia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Lazio
  - IRCCS Ospedale San Raffaele, Milan, Lombardy
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, Lombardy
  - Azienda Ospedaliera Universitaria Città della Salute e della Scienza di Torino, Turin, Piedmont
  - Università Politecnica delle Marche e AOU Ospedali Riuniti Umberto I°-Lancisi-Salesi , Ancona, Ancona, The Marches
  - ASL8 Arezzo San Donato Hospital, Arezzo, Tuscany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ammirati E, Frigerio M, Adler ED, Basso C, Birnie DH, Brambatti M, Friedrich MG, Klingel K, Lehtonen J, Moslehi JJ, Pedrotti P, Rimoldi OE, Schultheiss HP, Tschope C, Cooper LT Jr, Camici PG. Management of Acute Myocarditis and Chronic Inflammatory Cardiomyopathy: An Expert Consensus Document. Circ Heart Fail. 2020 Nov;13(11):e007405. doi: 10.1161/CIRCHEARTFAILURE.120.007405. Epub 2020 Nov 12. PMID 33176455
- [Background] Ammirati E, Raimondi F, Piriou N, Sardo Infirri L, Mohiddin SA, Mazzanti A, Shenoy C, Cavallari UA, Imazio M, Aquaro GD, Olivotto I, Pedrotti P, Sekhri N, Van de Heyning CM, Broeckx G, Peretto G, Guttmann O, Dellegrottaglie S, Scatteia A, Gentile P, Merlo M, Goldberg RI, Reyentovich A, Sciamanna C, Klaassen S, Poller W, Trankle CR, Abbate A, Keren A, Horowitz-Cederboim S, Cadrin-Tourigny J, Tadros R, Annoni GA, Bonoldi E, Toquet C, Marteau L, Probst V, Trochu JN, Kissopoulou A, Grosu A, Kukavica D, Trancuccio A, Gil C, Tini G, Pedrazzini M, Torchio M, Sinagra G, Gimeno JR, Bernasconi D, Valsecchi MG, Klingel K, Adler ED, Camici PG, Cooper LT Jr. Acute Myocarditis Associated With Desmosomal Gene Variants. JACC Heart Fail. 2022 Oct;10(10):714-727. doi: 10.1016/j.jchf.2022.06.013. Epub 2022 Sep 7. PMID 36175056
- [Background] Artico J, Merlo M, Delcaro G, Cannata A, Gentile P, De Angelis G, Paldino A, Bussani R, Ferro MD, Sinagra G. Lymphocytic Myocarditis: A Genetically Predisposed Disease? J Am Coll Cardiol. 2020 Jun 23;75(24):3098-3100. doi: 10.1016/j.jacc.2020.04.048. No abstract available. PMID 32553263
- [Background] Ammirati E, Moslehi JJ. Diagnosis and Treatment of Acute Myocarditis: A Review. JAMA. 2023 Apr 4;329(13):1098-1113. doi: 10.1001/jama.2023.3371. PMID 37014337
- [Background] Kontorovich AR, Patel N, Moscati A, Richter F, Peter I, Purevjav E, Selejan SR, Kindermann I, Towbin JA, Bohm M, Klingel K, Gelb BD. Myopathic Cardiac Genotypes Increase Risk for Myocarditis. JACC Basic Transl Sci. 2021 Jul 26;6(7):584-592. doi: 10.1016/j.jacbts.2021.06.001. eCollection 2021 Jul. PMID 34368507
- [Background] Lota AS, Hazebroek MR, Theotokis P, Wassall R, Salmi S, Halliday BP, Tayal U, Verdonschot J, Meena D, Owen R, de Marvao A, Iacob A, Yazdani M, Hammersley DJ, Jones RE, Wage R, Buchan R, Vivian F, Hafouda Y, Noseda M, Gregson J, Mittal T, Wong J, Robertus JL, Baksi AJ, Vassiliou V, Tzoulaki I, Pantazis A, Cleland JGF, Barton PJR, Cook SA, Pennell DJ, Garcia-Pavia P, Cooper LT Jr, Heymans S, Ware JS, Prasad SK. Genetic Architecture of Acute Myocarditis and the Overlap With Inherited Cardiomyopathy. Circulation. 2022 Oct 11;146(15):1123-1134. doi: 10.1161/CIRCULATIONAHA.121.058457. Epub 2022 Sep 26. PMID 36154167
- [Background] Lakkireddy D, Turagam MK, Yarlagadda B, Dar T, Hamblin M, Krause M, Parikh V, Bommana S, Atkins D, Di Biase L, Mohanty S, Rosamond T, Carroll H, Nydegger C, Wetzel L, Gopinathannair R, Natale A. Myocarditis Causing Premature Ventricular Contractions: Insights From the MAVERIC Registry. Circ Arrhythm Electrophysiol. 2019 Dec;12(12):e007520. doi: 10.1161/CIRCEP.119.007520. Epub 2019 Dec 16. PMID 31838913
- [Background] Tardif JC, Kouz S, Waters DD, Bertrand OF, Diaz R, Maggioni AP, Pinto FJ, Ibrahim R, Gamra H, Kiwan GS, Berry C, Lopez-Sendon J, Ostadal P, Koenig W, Angoulvant D, Gregoire JC, Lavoie MA, Dube MP, Rhainds D, Provencher M, Blondeau L, Orfanos A, L'Allier PL, Guertin MC, Roubille F. Efficacy and Safety of Low-Dose Colchicine after Myocardial Infarction. N Engl J Med. 2019 Dec 26;381(26):2497-2505. doi: 10.1056/NEJMoa1912388. Epub 2019 Nov 16. PMID 31733140
- [Background] Vandenburgh H, Shansky J, Benesch-Lee F, Barbata V, Reid J, Thorrez L, Valentini R, Crawford G. Drug-screening platform based on the contractility of tissue-engineered muscle. Muscle Nerve. 2008 Apr;37(4):438-47. doi: 10.1002/mus.20931. PMID 18236465
- [Background] Stoehr A, Neuber C, Baldauf C, Vollert I, Friedrich FW, Flenner F, Carrier L, Eder A, Schaaf S, Hirt MN, Aksehirlioglu B, Tong CW, Moretti A, Eschenhagen T, Hansen A. Automated analysis of contractile force and Ca2+ transients in engineered heart tissue. Am J Physiol Heart Circ Physiol. 2014 May;306(9):H1353-63. doi: 10.1152/ajpheart.00705.2013. Epub 2014 Feb 28. PMID 24585781